CLINICAL TRIAL: NCT02323451
Title: A Multicentre, Randomized, Double-blinded, Parallel-controlled, Non-inferiority Clinical Study Of Safety and Efficacy Of Medical Chitosan for Knee Osteoarthritis Compared With Sodium Hyaluronate Injection
Brief Title: Medical Chitosan or Sodium Hyaluronate for Knee Osteoarthritis (CHOOSE)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Qisheng Biological Preparation Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QS20140506
Record Dates: First submitted 2014-12-18; First posted 2014-12-23 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Medical Chitosan (Experimental): Medical Chitosan, 2ml/vial (12mg/ml), intra-articular injection with a volume less than 2ml every two weeks, a total of 3 times
  Interventions: Device: Medical Chitosan
- Sodium Hyaluronate Injection (Active Comparator): Sodium Hyaluronate Injection, 2ml/vial (10mg/ml), intra-articular injection with a volume less than 2ml every one weeks, a total of 5 times.
  Interventions: Drug: Sodium Hyaluronate Injection

INTERVENTIONS:
Device: Medical Chitosan — intra-articular injection
  Arms: Medical Chitosan
Drug: Sodium Hyaluronate Injection — intra-articular injection
  Arms: Sodium Hyaluronate Injection

SUMMARY:
This study evaluates the safety and efficacy of investigational products in the treatment of knee Osteoarthritis. Half of participants will receive medical chitosan, while the other half will receive sodium hyaluronate.

DETAILED DESCRIPTION:
Medical chitosan and sodium hyaluronate each form the reticular layer to cover the joint surface, alleviate the joint friction and pain. For medical chitosan, its half-life is longer than sodium hyaluronate, so the interval time of intra-articular injection is longer.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females at the age of 40-75 years old
2. Conforming to the diagnosis standard of the American College of Rheumatology in 2009： knee pain and osteophyte determined with X-ray, and at least one of the following items：

   * above 50 years old
   * morning stiffness less than 30 minutes
   * knee joint with fricative when moving
3. The studying knee has score of 40-90 mm on a 100 mm measured VAS and the other side was less than 40mm when walking on flat ground.
4. The studying knee has score of 1, 2 or 3 determined by radiological Kellgren-Lawrence grading scale.
5. Patients who have treatment requirements and can obey the therapeutic schedule
6. Body mass index(BMI) ≤35kg/m2。
7. Able to follow the clinical observation and follow up.
8. The subjects are able to understand and sign the informed consent after fully understand this study, the disease, investigational drugs, the therapeutic schedule and the potential risks.

Exclusion Criteria:

1. Positive signs of swelling or floating patella test，and there are obvious effusion of knee joint in clinical.
2. Other inflammatory pain diseases of knee joint, such as rheumatism/ rheumatoid arthritis, psoriatic arthritis, gout, hemophilic arthritis, etc.
3. Pain diseases of knee joint, except for osteoarthritis, such as intra-articular tumor, villonodular synovitis, joint trauma, etc.
4. Pregnant or lactating females.
5. Participants who suffer from serious cardiovascular disease (Sudden cerebral infarction with sequela or myocardial infarction within recent 6 months), hepatic disease, kidney disease；Participants whose ALT and AST are twice or more than twice than that of the upper limit of normal value；Participants whose serum creatinine exceed the upper limit of normal value；Participants who suffer from dysfunction of blood coagulation (thrombocytopenia, bleeder disease, etc.)
6. Participants who have systemic infection or infectious disease.
7. Participants who suffer from serious skin defect or ulcer around the studying knee joint.
8. Participants who suffer from typical varus or valgus deformities or lack of articular cavity.
9. Participants with diabetes and have to inject insulin or who are not good enough to control the blood glucose (FBG ( fasting blood-glucose) ≥10mmol/L.)
10. Participants who suffer from cancer (within 5 years) or Alzheimer's disease.
11. Participants with score 0 or 4 of the studying knee joint evaluated by radiological Kellgren-Lawrence grading scale.
12. Participants who have hormone drugs within 2 weeks or analgesic drugs within 1 week before this trial or take part in other clinical trials.
13. Participants whose studying knee receives articular cavity therapy within 3 months, containing intra articular administration, articular irrigation and arthroscopic surgery
14. Participants with an allergy to the experimental drugs.
15. Participants who are not suitable for this trial judged by the researchers.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-08 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale for knee pain | six weeks of the initial injection
  The investigator and the subject both evaluate the pain intensity per VAS before injection. VAS ranges from o to 10, 0=no pain, 10=pain as bad as can be.

SECONDARY OUTCOMES:
WOMAC for knee pain | six weeks of the initial injection
  WOMAC includes 3 items: pain, stiff and physiological function. 0=no, 4=as bad as can be.

CONTACTS AND LOCATIONS:
Overall Officials: Changqing Zhang, PhD, Principal Investigator — Shanghai,China.Shanghai Sixth People's Hospital. Orthopedics. Recruiting. No. 600. Yishan Rd. Shanghai. Post Code:200233.; Shigui Yan, PhD, Principal Investigator — Hangzhou,Chian. The Second Affiliated Hospital of Zhejiang University School of Medicine. Orthopedics. Not yet recruiting. No.88 Jiefang Road Hangzhou.China Post Code：310009
Locations (1):
- Shanghai Sixth People's Hospital. Orthopedics., Shanghai, Shanghai Municipality, China